CLINICAL TRIAL: NCT04207268
Title: Growing Healthy Hearts: A Pilot Randomized Control Trial to Test Gardening as an Intervention to Improve Dietary Intake of Fruits and Vegetables and Cardiovascular Disease Risk
Brief Title: Growing Healthy Hearts: A Pilot Randomized Control Trial to Test Gardening as an Intervention to Improve Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol could not be initiated due to COVID.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Susan Veldheer, Assistant Professor, Department of Family and Community Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00013976
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Gardening

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gardening and Nutrition Advice (Experimental): Participate in gardening activities, food demonstrations and nutrition advice
  Interventions: Behavioral: Gardening and Nutrition Advice
- Nutrition Advice alone (Placebo Comparator): Participate in only nutrition advice
  Interventions: Behavioral: Nutrition Advice

INTERVENTIONS:
Behavioral: Gardening and Nutrition Advice — Participate in gardening activities, gardening instructions and nutrition advice
  Arms: Gardening and Nutrition Advice
Behavioral: Nutrition Advice — Participate in only nutrition advice
  Arms: Nutrition Advice alone

SUMMARY:
The purpose of this study is to test the effect of group-based nutrition advice plus gardening (intervention) versus group-based nutrition advice alone on dietary intake of fruits and vegetables, physical activity, and lifetime risk for cardiovascular disease (CVD).

DETAILED DESCRIPTION:
Study participants will be randomly assigned to attend group sessions related to gardening with nutrition advice or nutrition advice alone. The main goal of the intervention will be to encourage participants to increase their intake of fruits and vegetables.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 20 years old
2. Have transportation and are willing to travel to the Hershey Community Garden
3. Have any two health conditions or risk factors for CVD. These include, but are not limited to:

   1. Any history of cardiovascular disease
   2. Any family history of premature cardiovascular disease
   3. Any history of stroke
   4. High cholesterol
   5. High blood pressure
   6. Overweight/obesity (BMI >=25)
   7. Diabetes
   8. Current or past Tobacco use

Exclusion Criteria:

1. Currently tends a vegetable garden
2. Moving out of the area in the next 4 months
3. Non-English speaking
4. Pregnant women
5. Participation in a past gardening study
6. Medical conditions or medications that limit ability to freely increase dietary intake of fruits and vegetables (e.g., kidney failure, dialysis)
7. A medical condition that precludes safe pursuit of gardening, i.e., recent heart conditions (e.g., heart failure, stroke, heart attack), recent or pending surgery, severe orthopedic conditions, pending hip/knee replacement, paralysis, dementia, blindness, unstable angina or uncontrolled arrhythmias, or uncontrolled asthma or allergies.
8. History of difficulty obtaining blood samples or fear of needles

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Plasma Carotenoids | 4 months
  The primary outcome is between group differences in total plasma carotenoids from baseline to 16 weeks. Plasma carotenoids are a reliable bio-marker of dietary intake of F&V.
Self-reported dietary intake | 4 months
  Investigators will also test the between group differences in self-reported servings of fruits and vegetables as assessed by 24-hour recalls.

SECONDARY OUTCOMES:
Cardiovascular disease risk score | 4 months
  Differences in Cardiovascular Disease (CVD) risk score based on the American College of Cardiology/American Heart Association (ACC/AHA) lifetime CVD risk score calculation (risk score range 0-100%). Higher scores indicate greater risk of a lifetime CVD-related event.
Physical activity | 4 months
  Between group differences in minutes of physical activity as measured by the International Physical Activity Questionnaire (IPAQ), (range in minutes, 0-3000+). Higher scores indicate more physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Veldheer, DEd, RD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No